CLINICAL TRIAL: NCT00255567
Title: A Multicentre Comparative Trial of Efficacy and Safety of Sodium Stibogluconate (SSG) Versus Paromomycin (PM) Versus Combination of SSG and PM as the First Line Treatment for Visceral Leishmaniasis in Ethiopia, Kenya and Sudan
Brief Title: Efficacy/Safety of Sodium Stibogluconate (SSG) Versus Paromomycin (PM) and SSG/PM Combination to Treat V Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-LEAP0104
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral Leishmaniasis; Combination
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Antimony Sodium Gluconate; Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Sodium Stibogluconate (30 days)
  Interventions: Drug: Sodium Stibogluconate
- 2 (Experimental): Paromomycin Sulphate (21 days)
  Interventions: Drug: Paromomycin sulphate
- 3 (Experimental): Sodium Stibogluconate + Paromomycin Sulphate (17 days)
  Interventions: Drug: SSG and Paromomycin sulphate

INTERVENTIONS:
Drug: Sodium Stibogluconate — Sodium Stibogluconate 20mg/kg/day for 30 days
  Arms: 1
Drug: Paromomycin sulphate — Paromomycin sulphate
  Arms: 2
Drug: SSG and Paromomycin sulphate — SSG and Paromomycin Sulphate 17 days
  Arms: 3

SUMMARY:
The purpose of this study is to assess the efficacy and safety of SSG 30 days alone, PM 21 days alone and SSG and PM as a combination course of 17 days in the treatment of patients with VL.

DETAILED DESCRIPTION:
Currently in the three countries, Sudan, Kenya and Ethiopia many of the patients present themselves in remote areas and need to be treated in relative resource poor settings. It is for this reason that standardised treatment with proven efficacy is much needed. A shorter course of treatment is not only advantageous for the patient but also reduces the overall case load in the clinics thus reducing the risk of disease outbreaks in already immuno-compromised kala-azar patients. Paromomycin, either alone or in combination with SSG would decrease the treatment duration substantially. An additional added value of combination therapy is that it is likely to reduce the chances of development of parasite resistance against the individual drugs.

Leishmaniasis experts in the three countries are in agreement that there are potential benefits of the combination treatment of SSG and PM and that its efficacy should be evaluated with the view to introduce this protocol if proven efficacious and safe. There is ample circumstantial evidence of the use of this combination therapy and its efficacy and tolerability as a standardized protocol. This can only be confirmed through a randomised controlled study with 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients for whom written informed consent has been signed by the patients themselves (if aged 18 years and over) or by parents(s) or legal guardian for patients under 18 years of age.
2. Patients aged between 4 and 60 years (inclusive) who are able to comply with the protocol. It is justified to include children because they represent more than 50% of VL cases.
3. Patients with clinical signs and symptoms of VL and diagnosis confirmed by visualization of parasites in tissue samples (spleen, lymph node or bone marrow) on microscopy.

Exclusion Criteria:

1. Patients who have received any anti-leishmanial drug in the last 6 months.
2. Patients with a negative splenic / lymph node / bone marrow smears.
3. Patients with a clinical contraindication to splenic/lymph node/ bone marrow aspirates.
4. Patients with severe protein and or caloric malnutrition (Kwashiokor or marasmus)
5. Patients with previous hypersensitivity reaction to SSG or aminoglycosides.
6. Patients suffering from a concomitant severe infection such as TB or any other serious underlying disease (cardiac, renal, hepatic) which would preclude evaluation of the patients response to study medication.
7. Patients suffering from other conditions associated with splenomegaly such as schistosomiasis.
8. Patients with previous history of cardiac arrhythmia or an abnormal ECG
9. Patients who are pregnant or lactating.
10. Patients with haemoglobin < 5gm/dl.
11. Patients with WBC < 1 x 10³/mm³.
12. Patients with platelets < 40,000/mm³.
13. Patients with liver function tests more than three times the normal range
14. Patients with serum creatinine outside the normal range for age and gender
15. Patients with pre-existing clinical hearing loss.

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1142 (Actual)
Dates: Start 2004-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
parasitological clearance at 6 months post treatment by splenic, lymph node, or bone marrow smear. | 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Manica Balasegaram, Study Director — Drugs for Neglected Diseases
Locations (5):
- Ethiopia (2):
  - Arba Minch Hospital, Arba Minch
  - Gondar hospital, Gonder
- KEMRI, Nairobi, Kenya
- Kassab Hospital, Kassāb, Sudan
- Amudat Hospital, Amudat, Nakipiripirit District, Uganda

REFERENCES:
- [Derived] Musa A, Khalil E, Hailu A, Olobo J, Balasegaram M, Omollo R, Edwards T, Rashid J, Mbui J, Musa B, Abuzaid AA, Ahmed O, Fadlalla A, El-Hassan A, Mueller M, Mucee G, Njoroge S, Manduku V, Mutuma G, Apadet L, Lodenyo H, Mutea D, Kirigi G, Yifru S, Mengistu G, Hurissa Z, Hailu W, Weldegebreal T, Tafes H, Mekonnen Y, Makonnen E, Ndegwa S, Sagaki P, Kimutai R, Kesusu J, Owiti R, Ellis S, Wasunna M. Sodium stibogluconate (SSG) & paromomycin combination compared to SSG for visceral leishmaniasis in East Africa: a randomised controlled trial. PLoS Negl Trop Dis. 2012;6(6):e1674. doi: 10.1371/journal.pntd.0001674. Epub 2012 Jun 19. PMID 22724029
- [Derived] Musa AM, Younis B, Fadlalla A, Royce C, Balasegaram M, Wasunna M, Hailu A, Edwards T, Omollo R, Mudawi M, Kokwaro G, El-Hassan A, Khalil E. Paromomycin for the treatment of visceral leishmaniasis in Sudan: a randomized, open-label, dose-finding study. PLoS Negl Trop Dis. 2010 Oct 26;4(10):e855. doi: 10.1371/journal.pntd.0000855. PMID 21049063